CLINICAL TRIAL: NCT03590730
Title: Benefits of ICD for the Primary Prevention in Patients With Valvular Cardiomyopathy
Acronym: BEAT
Status: Terminated | Type: Observational
Why Stopped: The trial stopped prematurely because of enrollment challenges.
Sponsor: Keimyung University Dongsan Medical Center (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor
Other Study IDs: 2017-08-027-007
Record Dates: First submitted 2018-07-02; First posted 2018-07-18 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2023-05

CONDITIONS: Valvular Heart Disease; Implantable Cardioverter Defibrillator; Sudden Cardiac Death; Primary Prevention
MeSH Terms: conditions — Heart Valve Diseases; Death, Sudden, Cardiac

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Valvular heart disease: Patients with left ventricular dysfunction due to valvular heart disease who received ICD implantation for primary prevention of sudden cardiac death.
  Interventions: Device: ICD implantation

INTERVENTIONS:
Device: ICD implantation — ICD will be implanted according to current guidelines recommendations.

SUMMARY:
The prevalence of valvular heart disease is on the rise along with the aging society and the generalization of echocardiography. Furthermore, the rheumatic valvular heart disease is much more prevalent in Asia than in Western countries, and the frequency of valve disease is higher in Asia. The effect of an implantable cardioverter defibrillator (ICD) in the primary prevention of sudden cardiac death in ischemic cardiomyopathy is well established and has become a standard of care. However, there is limited research on the effect of ICD implantation for primary prevention in patients with heart failure due to valvular heart disease. In a small study, the incidence of fatal cardiac arrhythmia was lower in patients with valvular cardiomyopathy (5%) who received ICD implantation for primary prevention than in those with ischemic cardiomyopathy. But there is also a report that the appropriate ICD treatment is not different from that of ischemic heart disease in valvular heart disease patients. Therefore, it is necessary to study the primary prevention effect of ICD on valvular cardiomyopathy in a larger number of patients. The purpose of this study was to investigate the effect of ICD on the prevention of sudden cardiac death in patients with heart failure due to valvular heart disease through prospective, multicenter, and observational studies.

ELIGIBILITY:
Inclusion Criteria:

* Patients who meet one of the following criteria:

  * Patients who have undergone surgery for aortic valve or mitral valve disease for more than 12 months
  * Patients with severe aortic valve or mitral valve disease
* Patients with left ventricular ejection fraction ≤ 35% by echocardiography or other imaging methods
* US, European practice guidelines class I indication for ICD implantation
* Patients without evidence of ischemic heart disease (who meet one of the following criteria):

  * Stress test negative
  * Significant stenosis was not observed in coronary artery images:

epicardial coronary stenosis <70%, left main stenosis <50%

* History of heart failure symptoms
* Patients who have received medication for more than 3 months according to the heart failure treatment guideline recommendation

Exclusion Criteria:

* Patients with left ventricular dysfunction without valvular heart disease
* Patients who require cardiac pacing therapy due to bradycardia
* Heart transplant scheduled
* Life expectancy is less than one year

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * South Korean patients visiting the one of the investigator's study participating hospital will be enrolled.
  * Valvular cardiomyopathy patients with left ventricular ejection fraction ≤ 35% with symptoms of NYHA class II, III despite optimal medical treatment for more than 3 months according to the guideline recommendations for heart failure treatment and are expected to survive for more than one year.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2017-11-15 (Actual); Primary Completion 2019-07-10 (Actual); Study Completion 2021-07-15 (Actual)

PRIMARY OUTCOMES:
Incidence of Appropriate ICD therapy | Two year after study enrollment
  ICD therapy that effectively terminate life-threatening arrhythmia: anti-tachycardia pacing, shock therapy

SECONDARY OUTCOMES:
Mortality | Two year after study enrollment
  mortality was recorded and it will be classified into cardiogenic/non-cardiogenic death. Especially, arrhythmic death was recorded separately.
Incidence of inappropriate ICD therapy | Two year after study enrollment
  Inappropriately delivered ICD therapy (eg. ICD therapy delivered during sinus tachycardia)
Type of ventricular arrhythmia | Two year after study enrollment
  Analyze the type of ventricular arrhythmia

CONTACTS AND LOCATIONS:
Overall Officials: Seongwook Han, MD, Ph D, Principal Investigator — Keimyung University Dongsan Medical Center
Locations (12):
- South Korea (12):
  - Pusan National University Yangsan Hospital, Yangsan, Gyeongsangnam-do
  - Division of Cardiology, Department of Internal Medicine, Kyungpook National University Hospital, Daegu
  - Division of Cardiology, Department of Internal Medicine, Yeungnam University Hospital, Daegu
  - Chonnam National University Hospital, Gwangju
  - Mediplex Sejong Hospital, Incheon
  - Seoul National University Bundang Hospital, Seongnam
  - Korea University Anam Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Cardiovascular Hospital, Seoul
  - Seoul Asan Medical Center, Seoul
  - Seoul Samsung Medical Center, Seoul
  - Seoul St. Mary's Hospital, Seoul

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for all primary and secondary outcome measures will be made available.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available within 6 months of study completion.
Access Criteria: Data access requests will be reviewed by an external independent Review Panel. Requestors will be required to sign a Data Access Agreement.